CLINICAL TRIAL: NCT00723450
Title: The Evaluation of Lamictal as an Add-on Treatment for Bipolar I Disorder in Children and Adolescents, 10 to 17 Years of Age
Brief Title: Lamictal as Add-on Treatment for Bipolar I Disorder in Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCA102833
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I pediatric lamictal adolescent
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Placebo Controlled
  Interventions: Drug: lamictal
- lamictal (Experimental): Flexible Dosing
  Interventions: Drug: lamictal

INTERVENTIONS:
Drug: lamictal — Flexible Dosing

SUMMARY:
The study will be a multi-center, parallel, group, placebo control, double-blind, randomized controlled trial of lamictal as add-on maintenance treatment in pediatric outpatients (aged 10 to 17 years) diagnosed with Bipolar I disorder. The study consists of 4 phases: Screen (approximately 2 weeks), Open label phase (up to 18 weeks), Randomized phase (up to 36 weeks) and Taper and follow-up phase (up to 4 weeks).

ELIGIBILITY:
Inclusion Criteria

* Subject is male or female between the ages of 10 and 17 years, inclusive.
* Subject has a diagnosis of bipolar I disorder and is currently experiencing a manic/hypomanic, depressed, or mixed mood episode
* Subject is currently receiving a stable treatment regimen.
* Subject is living with his/her custodial parent(s) or legal guardian(s) and has contact with them on a daily basis.

Exclusion Criteria

* Subject has been diagnosed with a primary Axis I disorder (with the exception of bipolar I disorder, ADHD, anxiety disorders, oppositional defiant disorder, or conduct disorder) or any Axis II disorder.
* Subject currently has signs or symptoms of psychosis or a history of psychosis within the previous four weeks.
* Subject has been diagnosed with epilepsy, autism, Asperger's syndrome, or Tourette's syndrome.
* Subject has experienced a serious rash, such as Stevens-Johnson Syndrome or Toxic Epidermal Necrolysis, or a rash otherwise requiring hospitalization.
* Subject has experienced a rash related to prior LAMICTAL use, or for whom LAMICTAL treatment was discontinued for clinically significant safety reasons.
* Subject has received any antidepressant medication, or atomoxetine, during the four weeks prior to the Screen Visit.
* Subject has initiated psychotherapy within 2 months prior to the Screen Visit, or plans to initiate psychotherapy during the trial.
* Subject in the 10-12 year old age group has a Body Mass Index (BMI) less than or equal 15 or greater than or equal to 30; a subject in the 13-17 year old age group has a BMI less than or equal to 17 or greater than or equal to 34.
* Subject tests positive for illicit drug use at the Screen Visit, has a history of alcohol or substance abuse or dependence (other than nicotine dependence) within the past three months, or has a positive blood alcohol level at the Screen Visit.
* Subject, in the investigator's judgment, poses a current homicidal or serious suicidal risk, has made a suicide attempt within the twelve months preceding the Screen Visit, has ever been homicidal.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 301 (Actual)
Dates: Start 2008-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (42):
- United States (42):
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Bradenton, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Smyrna, Georgia
  - GSK Investigational Site, Libertyville, Illinois
  - GSK Investigational Site, Naperville, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Piscataway, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Mount Kisco, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Roanoke, Virginia
  - GSK Investigational Site, Kirkland, Washington
  - GSK Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Findling RL, Chang K, Robb A, Foster VJ, Horrigan J, Krishen A, Wamil A, Kraus JE, DelBello M. Adjunctive Maintenance Lamotrigine for Pediatric Bipolar I Disorder: A Placebo-Controlled, Randomized Withdrawal Study. J Am Acad Child Adolesc Psychiatry. 2015 Dec;54(12):1020-1031.e3. doi: 10.1016/j.jaac.2015.09.017. Epub 2015 Oct 14. PMID 26598477
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: SCA102833 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SCA102833 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SCA102833 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SCA102833 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SCA102833 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SCA102833 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SCA102833 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 301 participants were enrolled in the study, of which 298 subjects took at least one dose of lamotrigine (LTG). One hundred and seventy three participants met stabilization criteria and entered the Randomized Phase.
Pre-assignment Details: The study consisted of a 2-week Screening Phase, an 18-week Open-Label Phase, a 36-week Double-Blind Randomized Phase and a Taper and Follow-up Phase (up to 4 weeks depending on the dose the participant was taking at the last Open-Label or Randomized Phase visit), which was either open-label or double-blind depending on the phase of the study.
Groups:
- LTG: Open-Label Phase: Participants (par.) received lamotrigine (LTG) up to a maximum dose depending on their age and concomitant bipolar medication group. Participants 10 -12 years of age received LTG up to a maximum dose of: 3 milligrams/kilograms (mg/kg)/day or 100 mg/day, whichever was less; or 6 mg/kg/day or 200 mg/day whichever was less; or 12 mg/kg/day or 300 mg/day whichever was less, depending on their bipolar medication group. Participants 13-17 years of age received LTG up to a maximum dose of 150 mg/day, 300 mg/day, or 400 mg/day depending on their bipolar medication group. Participants took LTG for a duration of up to 18 weeks.
- Placebo: Participants received matching placebo in the evening for participants taking one dose and for participants taking two divided doses, one dose in the morning and one dose in the evening, for a duration of up to 36 weeks.
- Lamotrigine: Participants received LTG equivalent to the dose established in the Open-Label Phase. Participants received LTG tablets in the evening for participants taking one dose and for participants taking two divided doses, one dose in the morning and one dose in the evening, for a duration of up to 36 weeks.
Period: Open-Label Phase
Arm/Group | LTG: Open-Label Phase | Placebo | Lamotrigine
Started | 298 | 0 | 0
Completed | 173 | 0 | 0
Not Completed | 125 | 0 | 0
Not completed — Adverse Event | 26 | 0 | 0
Not completed — Lack of Efficacy | 18 | 0 | 0
Not completed — Protocol Violation | 35 | 0 | 0
Not completed — Lost to Follow-up | 7 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Withdrawal by Subject | 37 | 0 | 0
Period: Randomized Phase
Arm/Group | LTG: Open-Label Phase | Placebo | Lamotrigine
Started | 0 | 86 | 87
Completed | 0 | 21 | 20
Not Completed | 0 | 65 | 67
Not completed — Adverse Event | 0 | 26 | 17
Not completed — Lack of Efficacy | 0 | 11 | 11
Not completed — Protocol Violation | 0 | 9 | 13
Not completed — Lost to Follow-up | 0 | 2 | 3
Not completed — Physician Decision | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 14 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lamotrigine | Total
Number analyzed (Participants) | 86 | 87 | 173
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.5 (2.22) | 13.4 (2.33) | 13.5 (2.27)
Gender [Count of Participants; unit: Participants]
  Female | 39 | 33 | 72
  Male | 47 | 54 | 101
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 9 | 9 | 18
  American Indian or Alaska Native | 0 | 1 | 1
  Asian - East Asian Heritage | 1 | 0 | 1
  White - Arabic/North African Heritage | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 71 | 71 | 142
  Mixed Race | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to the Occurrence of a Bipolar Event (TOBE)
Description: TOBE was defined by the first prescription of any additional pharmacotherapy to treat bipolar symptoms, increasing the dose(s) of the participants conventional bipolar medication(s), treatment with electroconvulsive therapy, or moving the participant to a more restricted environment for observation, safety, or treatment; or participant withdrawal from the study due to a bipolar-related adverse event (AE) or serious adverse event (SAE); or participants withdrawal from the study due to lack of efficacy as defined by rating scale threshold scores. TOBE was calculated using a log rank test with stratification for index mood state (depression, mania/hypomania, mixed mood).
Time Frame: From randomization until Week 36
Population: Randomized Intent-to-Treat (ITT) Population: all participants who were randomized to LTG or placebo and received at least one dose of investigational product.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 86 | 87
Days
  Stratum: Depression, n=22,21 | 50 (3.8) | 155 (14.7)
  Stratum: Mania/Hypomania, n=36, 37 | 120 (12.2) | 163 (12.2)
  Stratum: Mixed Mood, n=28, 29 | 107 (13.8) | 136 (15.4)
Statistical Analysis 1: Comparison: Placebo vs Lamotrigine; Test type: Superiority or Other; p = 0.0717, Log Rank; A stratified log rank test was performed where the stratification factor was the index mood state at Screen visit

2. Secondary Outcome: Time From Randomization to Withdrawal From the Study for Any Cause (TTW)
Description: The time from randomization to the withdrawal from study was analyzed. TTW was calculated using the log rank test with stratification for index mood state (depression, mania/hypomania, mixed mood).
Time Frame: From randomization until withdrawal from the study for any cause (up to Week 36)
Population: Randomized ITT Population
Measure: Mean (Standard Error); unit: Days
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 86 | 87
Days
  Stratum: Depression, n=22, 21 | 113 (21.4) | 141 (20.0)
  Stratum: Mania/Hypomania, n=36, 37 | 138 (17.3) | 144 (15.6)
  Stratum: Mixed Mood, n=28, 29 | 101 (15.7) | 106 (16.3)

3. Secondary Outcome: Time From Randomization to Intervention for a Mood Episode (TIME)
Description: The time from randomization to the intervention for a mood episode (depression, mania/hypomania or mixed mood) was analyzed. TIME was calculated using the log rank test with stratification for index mood state (depression, mania/hypomania, mixed mood).
Time Frame: From randomization until intervention administered for a mood episode (up to Week 36)
Population: Randomized ITT Population
Measure: Mean (Standard Error); unit: Days
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 86 | 87
Days
  Stratum: Depression, n=22, 21 | 62 (5.2) | 164 (12.7)
  Stratum: Mania/Hypomania, n=36, 37 | 129 (11.7) | 179 (10.8)
  Stratum: Mixed Mood, n=28, 29 | 120 (13.7) | 127 (12.0)

4. Secondary Outcome: Time From Randomization to Intervention for Depression (TIDep), Mania/Hypomania (TIMan), or a Mixed Episode (TIMix)
Description: The time from randomization to intervention for depression (TIDep), mania/hypomania (TIMan), or a mixed episode (TIMix) was analyzed. TIDep, TIMan, and TIMix were calculated using the log rank test with stratification for index mood state (depression, mania/hypomania, mixed mood).
Time Frame: From randomization until intervention administered for depression, mania/hypomania or a mixed episode (up to Week 36)
Population: Randomized ITT Population
Measure: Mean (Standard Error); unit: Days
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 86 | 87
Days
  TIDep: Depression, n=22, 21 | 61 (1.5) | 46 (1.5)
  TIDep: Mania/Hypomania, n=36, 37 | NA (NA) — There were zero events for this endpoint in this stratum, therefore, the mean and the standard error could not be estimated. | NA (NA) — There were zero events for this endpoint in this stratum, therefore, the mean and the standard error could not be estimated.
  TIDep: Mixed Mood, n=28, 29 | 59 (2.6) | 159 (NA) — There were 0-1 events for this endpoint in this stratum, therefore, the standard error could not be estimated.
  TIMan: Depression, n=22, 21 | 74 (3.9) | 182 (NA) — There were 0-1 events for this endpoint in this stratum, therefore, the standard error could not be estimated.
  TIMan: Mania/Hypomania, n=36, 37 | 139 (11.5) | 61 (2.1)
  TIMan: Mixed Mood, n=28, 29 | 105 (7.3) | 148 (8.5)
  TIMix: Depression, n=22, 21 | 37 (1.3) | 158 (NA) — There were 0-1 events for this endpoint in this stratum, therefore, the standard error could not be estimated.
  TIMix: Mania/Hypomania, n=36, 37 | 135 (6.3) | 194 (7.5)
  TIMix: Mixed Mood, n=28, 29 | 160 (10.7) | 57 (2.5)

5. Secondary Outcome: Number of Participants Experiencing a Relapse/Recurrence to Depression, Mania/Hypomania, or Mixed Mood State
Description: The number of participants requiring intervention to treat either the emergence of or a change in bipolar symptoms that is, experiencing a relapse/recurrence to depression, mania/hypomania, or mixed mood state were analyzed.
Time Frame: From randomization until a relapse/recurrence to depression, mania/hypomania, or mixed mood state (up to Week 36)
Population: Randomized ITT Population. Only those participants requiring intervention to treat either the emergence of, or a change, in bipolar symptoms were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 31 | 18
Participants
  Depression | 5 | 3
  Mania/hypomania | 16 | 6
  Mixed episode state | 10 | 9

6. Secondary Outcome: Number of Participants Experiencing a Relapse/Recurrence Within the First 30, 90, and 180 Days in the Randomized Phase
Description: The proportion of participants (par.) requiring intervention to treat either the emergence of or a change in bipolar symptoms, that is, experiencing a relapse/recurrence to depression, mania/hypomania, or mixed mood state at any time within the first 30, 90, and 180 days in the Randomized Phase were analyzed.
Time Frame: From randomization up to Week 36
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 31 | 18
Participants
  Mania/hypomania, 30 days, n=16, 6 | 9 | 2
  Mania/hypomania, 90 days, n=16, 6 | 12 | 4
  Mania/hypomania, 180 days, n=16, 6 | 16 | 5
  Depression, 30 days, n=5, 3 | 1 | 1
  Depression, 90 days, n=5, 3 | 5 | 2
  Depression, 180 days, n=5, 3 | 5 | 3
  Mixed mood state, 30 days, n= 10, 9 | 3 | 2
  Mixed mood state, 90 days, n= 10, 9 | 7 | 6
  Mixed mood state, 180 days, n= 10, 9 | 10 | 8

7. Secondary Outcome: Change From Baseline in the Quick Inventory of Depressive Symptomatology - Clinician Interview, Semi-structured, Adolescent Version (QIDS- A17-C) at Each Visit in the Open-Label Phase
Description: The QIDS-A17-C is a 17-item scale used to assess depression severity in adolescents according to the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) diagnostic criteria for a major depressive episode; it is a modified version of the Quick Inventory of Depressive Symptomatology (QIDS) used for adults. Each item is scored on a 0-3 scale, yielding 9 domain scores. The range of scores is 0 (best possible outcome) to 27 (worst possible outcome). Analysis was performed using mixed model repeated measures.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, and 18
Population: Open-Label ITT population: all participants who entered the Open-Label Phase and received at least one dose of LTG.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Groups:
- LTG: Open-Label Phase: Participants (par.) received lamotrigine (LTG) up to a maximum dose depending on their age and concomitant bipolar medication group. Participants 10 -12 years of age received LTG up to a maximum dose of : 3 milligrams/kilograms (mg/kg)/day or 100 mg/day, whichever was less; or 6 mg/kg/day or 200 mg/day whichever was less; or 12 mg/kg/day or 300 mg/day whichever was less, depending on their bipolar medication group. Participants 13-17 years of age received LTG up to a maximum dose of 150 mg/day, 300 mg/day, or 400 mg/day depending on their bipolar medication group. Participants took LTG for a duration of up to 18 weeks.
Arm/Group | LTG: Open-Label Phase
Number analyzed (Participants) | 298
Scores on a Scale
  Week 1 | -2.1 (0.22)
  Week 2 | -2.9 (0.28)
  Week 3 | -3.7 (0.28)
  Week 4 | -3.8 (0.30)
  Week 5 | -4.3 (0.30)
  Week 6 | -4.7 (0.30)
  Week 7 | -5.1 (0.30)
  Week 8 | -4.9 (0.31)
  Week 9 | -5.6 (0.30)
  Week 10 | -6.1 (0.29)
  Week 11 | -6.4 (0.30)
  Week 12 | -6.6 (0.32)
  Week 13 | -6.7 (0.32)
  Week 14 | -6.8 (0.34)
  Week 15 | -6.8 (0.40)
  Week 16 | -6.8 (0.41)
  Week 17 | -6.5 (0.53)
  Week 18 | -6.5 (0.70)

8. Secondary Outcome: Change From Randomization in the Quick Inventory of Depressive Symptomatology - Clinician Interview, Semi-structured, Adolescent Version (QIDS- A17-C) at Each Visit in the Randomized Phase
Description: as for outcome 7
Time Frame: Randomization and Weeks 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, and 36
Population: Randomized ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 86 | 87
Scores on a scale
  Week 1 | 0.8 (0.30) | 0.5 (0.31)
  Week 2 | 1.5 (0.37) | 1.1 (0.37)
  Week 3 | 1.3 (0.36) | 0.6 (0.36)
  Week 4 | 1.2 (0.39) | 1.0 (0.39)
  Week 6 | 1.9 (0.49) | 1.5 (0.47)
  Week 8 | 1.9 (0.47) | 1.7 (0.45)
  Week 10 | 1.4 (0.44) | 1.5 (0.41)
  Week 12 | 1.4 (0.40) | 1.2 (0.39)
  Week 16 | 2.2 (0.48) | 1.8 (0.47)
  Week 20 | 1.5 (0.50) | 2.5 (0.46)
  Week 24 | 1.7 (0.53) | 1.8 (0.51)
  Week 28 | 1.6 (0.61) | 2.3 (0.57)
  Week 32 | 1.0 (0.72) | 1.9 (0.72)
  Week 36 | 2.3 (0.63) | 1.9 (0.63)

9. Secondary Outcome: Change From Baseline in the Quick Inventory of Depressive Symptomatology - Self-report Adolescent Version (QIDS-A17-SR) at Each Visit in the Open-Label Phase
Description: The QIDS-A17-SR is a 17-item scale used to assess depression severity in adolescents according to the DSM-IV-TR diagnostic criteria for a major depressive episode; it is a modified version of the Quick Inventory of Depressive Symptomatology (QIDS) used for adults. Each item is scored on a 0-3 scale, yielding 9 domain scores. The range of scores is 0 (best possible outcome) to 27 (worst possible outcome). The scale is completed by the participant. Analysis was performed using mixed model repeated measures.
Time Frame: Baseline and Weeks 4, 8, 12, 16, and 18
Population: Open-Label ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | LTG: Open-Label Phase
Number analyzed (Participants) | 298
Scores on a scale
  Week 4 | -2.7 (0.25)
  Week 8 | -3.3 (0.27)
  Week 12 | -4.3 (0.28)
  Week 16 | -4.5 (0.33)
  Week 18 | -5.0 (0.52)

10. Secondary Outcome: Change From Randomization in the Quick Inventory of Depressive Symptomatology - Self-report Adolescent Version (QIDS-A17-SR) at Each Visit in the Randomized Phase
Description: as for outcome 9
Time Frame: Randomization and Weeks 8, 16, 24, 32, and 36
Population: Randomized ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 86 | 87
Scores on a scale
  Week 8 | 1.6 (0.47) | 1.2 (0.48)
  Week 16 | 1.6 (0.60) | 1.4 (0.58)
  Week 24 | 1.0 (0.60) | 1.5 (0.56)
  Week 32 | 0.6 (0.66) | 0.2 (0.63)
  Week 36 | 0.9 (0.66) | 0.8 (0.68)

11. Secondary Outcome: Change From Baseline in the Clinical Global Impressions - Bipolar, Severity of Illness (CGI-BP[S]) at Each Visit in the Open-Label Phase
Description: Severity of the bipolar illness was based on the CGI-BP(S) score which had a range from 1 (normal, not ill) to 7 (very severely ill). Analysis was performed using mixed model repeated measures.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, and 18
Population: Open-Label ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | LTG: Open-Label Phase
Number analyzed (Participants) | 298
Scores on a scale
  Week 1 | -0.4 (0.05)
  Week 2 | -0.6 (0.05)
  Week 3 | -0.9 (0.06)
  Week 4 | -1.0 (0.06)
  Week 5 | -1.2 (0.06)
  Week 6 | -1.3 (0.06)
  Week 7 | -1.4 (0.07)
  Week 8 | -1.5 (0.07)
  Week 9 | -1.6 (0.07)
  Week 10 | -1.8 (0.07)
  Week 11 | -1.9 (0.07)
  Week 12 | -2.1 (0.07)
  Week 13 | -2.1 (0.07)
  Week 14 | -2.1 (0.07)
  Week 15 | -2.1 (0.08)
  Week 16 | -2.1 (0.10)
  Week 17 | -2.0 (0.12)
  Week 18 | -2.1 (0.15)

12. Secondary Outcome: Change From Randomization in the Clinical Global Impressions - Bipolar, Severity of Illness (CGI-BP[S]) at Each Visit in the Randomized Phase
Description: as for outcome 11
Time Frame: Randomization and Weeks 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, and 36
Population: Randomized ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 86 | 87
Scores on a scale
  Week 1 | 0.2 (0.09) | 0.0 (0.09)
  Week 2 | 0.4 (0.12) | 0.2 (0.12)
  Week 3 | 0.4 (0.12) | 0.2 (0.12)
  Week 4 | 0.6 (0.13) | 0.3 (0.13)
  Week 6 | 0.8 (0.15) | 0.4 (0.15)
  Week 8 | 0.7 (0.15) | 0.4 (0.14)
  Week 10 | 0.4 (0.13) | 0.6 (0.13)
  Week 12 | 0.5 (0.14) | 0.4 (0.14)
  Week 16 | 0.6 (0.17) | 0.6 (0.15)
  Week 20 | 0.5 (0.17) | 0.8 (0.16)
  Week 24 | 0.4 (0.17) | 0.6 (0.16)
  Week 28 | 0.3 (0.17) | 0.5 (0.16)
  Week 32 | 0.2 (0.19) | 0.5 (0.20)
  Week 36 | 0.4 (0.19) | 0.3 (0.21)

13. Secondary Outcome: Summary of Clinical Global Impressions - Bipolar - Improvement of Illness (CGI-BP [I]) Scores During Open-label Phase
Description: Improvement of bipolar illness was based on the CGI-BP (I) score which ranged from 1 (very much improved) to 7 (very much worse). Analysis was performed using mixed model repeated measures.
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, and 18
Population: Open-Label ITT Population. Only those par. available at the specified time points were analyzed (represented by n=X). Different par. may have been analyzed at different time points, so the overall number of par. analyzed reflects everyone in the Open-Label Population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LTG: Open-Label Phase
Number analyzed (Participants) | 298
Scores on a scale
  Week 1, n=290 | 3.6 (0.80)
  Week 2, n=278 | 3.3 (0.90)
  Week 3, n=270 | 3.1 (0.96)
  Week 4, n=265 | 3.0 (1.03)
  Week 5, n=258 | 2.8 (1.01)
  Week 6, n=243 | 2.7 (1.05)
  Week 7, n=246 | 2.5 (1.07)
  Week 8, n=236 | 2.5 (1.09)
  Week 9, n=227 | 2.3 (1.05)
  Week 10, n=205 | 2.2 (1.09)
  Week 11, n=181 | 2.2 (0.92)
  Week 12, n=168 | 2.0 (0.87)
  Week 13, n=141 | 1.9 (0.85)
  Week 14, n=118 | 1.9 (0.69)
  Week 15, n=93 | 1.8 (0.71)
  Week 16, n=72 | 2.0 (0.89)
  Week 17, n=42 | 2.0 (0.70)
  Week 18, n=28 | 2.0 (0.88)

14. Secondary Outcome: Summary of Clinical Global Impressions - Bipolar - Improvement of Illness (CGI-BP [I]) Scores During Randomized Phase
Description: Improvement of bipolar illness was based on the CGI-BP(I) score which ranged from 1 (very much improved) to 7 (very much worse). Analysis was performed using mixed model repeated measures.
Time Frame: Randomization weeks 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32 and 36
Population: Randomized ITT Population. Only those par. available at the specified time points were analyzed (represented by n=X). Different par. may have been analyzed at different time points, so the overall number of par. analyzed reflects everyone in the Randomized ITT Population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 86 | 87
Scores on a scale
  Week 1, n=84, 85 | 3.3 (1.40) | 3.3 (1.37)
  Week 2, n=82, 81 | 3.7 (1.48) | 3.6 (1.38)
  Week 3, n=74, 75 | 3.6 (1.39) | 3.6 (1.34)
  Week 4, n=65, 70 | 3.6 (1.51) | 3.6 (1.35)
  Week 6, n=58, 64 | 3.8 (1.64) | 3.4 (1.49)
  Week 8, n=51, 60 | 3.5 (1.72) | 3.6 (1.47)
  Week 10, n=45, 55 | 3.3 (1.64) | 3.8 (1.19)
  Week 12, n=45, 49 | 3.3 (1.52) | 3.4 (1.29)
  Week 16, n=43, 50 | 3.4 (1.73) | 3.5 (1.37)
  Week 20, n=37, 43 | 3.0 (1.48) | 3.8 (1.36)
  Week 24, n=34, 36 | 3.0 (1.59) | 3.4 (1.44)
  Week 28, n=29, 32 | 2.7 (1.56) | 3.5 (1.44)
  Week 32, n=28, 27 | 3.0 (1.63) | 3.5 (1.28)
  Week 36, n=27, 24 | 3.0 (1.68) | 3.6 (1.10)

15. Secondary Outcome: Number of Participants Considered Much Improved or Very Much Improved [Defined as a Clinical Global Impression-Bipolar Version, Improvement of Illness (CGI-BP[I]), Score of 1 or 2] at Each Visit Compared to Baseline in the Open-Label Phase
Description: The CGI-BP(I) asks the following question: "Compared to the Baseline assessment in this trial, how much has the participant changed?". Scores on the CGI-I range from 1 (very much improved) to 7 (very much worse). The investigator or their designee rated improvement regardless of whether the improvement to be due to drug treatment. Improvement defined as CGI-BP(I)=1 (improved) or 2 (very much improved). Missing data imputed using last-observation carried forward (LOCF).
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, and 18
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | LTG: Open-Label Phase
Number analyzed (Participants) | 298
Participants
  Week 1, n=297 | 27
  Week 2, n=297 | 46
  Week 3, n=297 | 72
  Week 4, n=297 | 86
  Week 5, n=297 | 113
  Week 6, n=297 | 124
  Week 7, n=297 | 138
  Week 8, n=297 | 140
  Week 9, n=297 | 159
  Week 10, n=297 | 176
  Week 11, n=297 | 182
  Week 12, n=297 | 195
  Week 13, n=297 | 205
  Week 14, n=297 | 211
  Week 15, n=297 | 210
  Week 16, n=297 | 209
  Week 17, n=297 | 208
  Week 18, n=297 | 206

16. Secondary Outcome: Number of Participants Considered Much Improved or Very Much Improved [Defined as a Clinical Global Impression-Bipolar Version, Improvement of Illness (CGI-BP[I]), Score of 1 or 2] at Each Visit Compared to Randomization in the Randomized Phase
Description: The CGI-BP(I) asks the following question: "Compared to the Randomization assessment in this trial, how much has the participant changed?". Scores on the CGI-I range from 1 (very much improved) to 7 (very much worse). The investigator or their designee rated improvement regardless of whether the improvement to be due to drug treatment. Improvement defined as CGI-BP(I)=1 (improved) or 2 (very much improved). Missing data imputed using last-observation carried forward (LOCF).
Time Frame: Randomization and Weeks 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, and 36
Population: Randomized ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 86 | 87
Participants
  Week 1 | 31 | 31
  Week 2 | 25 | 22
  Week 3 | 24 | 21
  Week 4 | 22 | 19
  Week 6 | 20 | 23
  Week 8 | 22 | 19
  Week 10 | 22 | 12
  Week 12 | 21 | 17
  Week 16 | 21 | 16
  Week 20 | 21 | 14
  Week 24 | 21 | 15
  Week 28 | 22 | 15
  Week 32 | 19 | 15
  Week 36 | 20 | 13

17. Secondary Outcome: Change From Baseline in the Young Mania Rating Scale (YMRS) at Each Visit in the Open-Label Phase
Description: The YMRS consists of 11 items and is based on the participant's report of their mania symptoms. It is clinician rated. Four items (irritability, speech, thought content, and disruptive/aggressive behavior) are rated on a scale of 0 to 8, while the other seven items (elevated mood, increased motor activity-energy, sexual interest, sleep, language, appearance, and insight) are rated on a scale of 0 to 4. The range of scores for the YMRS is 0 (best possible outcome) to 60 (worst possible outcome). The YMRS was completed by the investigator or their qualified designee. Analysis was performed using mixed model repeated measures.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, and 18
Population: Open-Label ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | LTG: Open-Label Phase
Number analyzed (Participants) | 298
Scores on a scale
  Week 1 | -3.2 (0.39)
  Week 2 | -4.8 (0.42)
  Week 3 | -6.4 (0.45)
  Week 4 | -6.5 (0.46)
  Week 5 | -7.5 (0.50)
  Week 6 | -8.4 (0.50)
  Week 7 | -9.1 (0.51)
  Week 8 | -8.8 (0.48)
  Week 9 | -9.6 (0.48)
  Week 10 | -10.3 (0.49)
  Week 11 | -11.1 (0.48)
  Week 12 | -11.6 (0.53)
  Week 13 | -12.0 (0.58)
  Week 14 | -12.0 (0.59)
  Week 15 | -12.4 (0.63)
  Week 16 | -12.3 (0.78)
  Week 17 | -12.2 (0.88)
  Week 18 | -12.1 (1.43)

18. Secondary Outcome: Change From Randomization in the Young Mania Rating Scale (YMRS) at Each Visit in the Randomized Phase
Description: as for outcome 17
Time Frame: Randomization and Weeks 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, and 36
Population: Randomized ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 86 | 87
Scores on a scale
  Week 1 | 1.3 (0.57) | 0.4 (0.59)
  Week 2 | 2.6 (0.72) | 2.1 (0.72)
  Week 3 | 2.6 (0.69) | 1.3 (0.71)
  Week 4 | 3.7 (0.85) | 2.0 (0.84)
  Week 6 | 4.9 (0.96) | 2.3 (0.93)
  Week 8 | 4.3 (0.98) | 3.5 (0.93)
  Week 10 | 3.5 (0.87) | 2.9 (0.82)
  Week 12 | 3.2 (0.84) | 1.6 (0.81)
  Week 16 | 4.7 (0.93) | 3.0 (0.89)
  Week 20 | 4.8 (0.99) | 4.5 (0.92)
  Week 24 | 4.2 (1.06) | 2.9 (1.02)
  Week 28 | 4.4 (1.04) | 3.7 (1.01)
  Week 32 | 4.5 (1.10) | 2.6 (1.14)
  Week 36 | 3.5 (0.92) | 1.2 (0.95)

19. Secondary Outcome: Change From Baseline in the Parent Version of the Young Mania Rating Scale (P-YMRS) at Each Visit in the Open-Label Phase
Description: The P-YMRS was adapted from the YMRS for completion by parents of the pediatric participants with bipolar disorder in order to assess the severity of the manic symptoms. The P-YMRS consisted of 11 items and had a total score range of 0 (best possible outcome) to 60 (worst possible outcome). The P-YMRS was completed by the participant's custodial parent or legal guardian. Analysis was performed using mixed model repeated measures.
Time Frame: Baseline and Weeks 4, 8, 12, 16, and 18
Population: Open-Label ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | LTG: Open-Label Phase
Number analyzed (Participants) | 298
Scores on a scale
  Week 4 | -4.7 (0.57)
  Week 8 | -6.0 (0.62)
  Week 12 | -7.4 (0.62)
  Week 16 | -8.2 (0.72)
  Week 18 | -9.3 (1.29)

20. Secondary Outcome: Change From Randomization in the Parent Version of the Young Mania Rating Scale (P-YMRS) at Each Visit in the Randomized Phase
Description: as for outcome 19
Time Frame: Randomization and Weeks 8, 16, 24, 32, and 36
Population: Randomized ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 86 | 87
Scores on a scale
  Week 8 | 4.9 (0.93) | 4.3 (0.95)
  Week 16 | 2.7 (1.13) | 2.6 (1.09)
  Week 24 | 5.3 (1.35) | 5.7 (1.29)
  Week 32 | 5.1 (1.33) | 6.0 (1.32)
  Week 36 | 5.3 (1.33) | 4.5 (1.36)

21. Secondary Outcome: Change From Baseline in the Conners' Global Index - Parent Version (CGI-P) at Each Visit in the Open-Label Phase
Description: The CGI-P is a 10-item scale used to assess attention deficit hyperactivity disorder (ADHD) symptoms in children and adolescents aged 3-17 years of age. The scale is composed of two factors: restless-impulsive behavior and emotional lability. Each item was scored on a 0-3 scale. The range of scores for the CGI-P is 0 (best possible outcome) to 30 (worst possible outcome). The CGI-P was completed by the participant's custodial parent or legal guardian. Analysis was performed using mixed model repeated measures.
Time Frame: Baseline and Weeks 4, 8, 12, 16, and 18
Population: Open-Label ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | LTG: Open-Label Phase
Number analyzed (Participants) | 298
Scores on a scale
  Week 4 | -4.0 (0.36)
  Week 8 | -5.7 (0.43)
  Week 12 | -6.7 (0.47)
  Week 16 | -7.1 (0.56)
  Week 18 | -8.2 (1.07)

22. Secondary Outcome: Change From Randomization in the Conners' Global Index - Parent Version (CGI-P) at Each Visit in the Randomized Phase.
Description: as for outcome 21
Time Frame: Randomization and Weeks 8, 16, 24, 32, and 36
Population: Randomized ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 86 | 87
Scores on a scale
  Week 8 | 3.1 (0.75) | 2.1 (0.77)
  Week 16 | 3.4 (0.92) | 1.2 (0.90)
  Week 24 | 2.4 (1.12) | 3.1 (1.05)
  Week 32 | 2.7 (1.10) | 2.6 (1.08)
  Week 36 | 1.5 (1.00) | 0.5 (1.03)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the first dose of investigational product until the last visit of the Open-Label or Double-Blind Taper and Follow-up Phase (up to Taper Week 4).
Description: On-treatment SAEs and non-serious AEs, were reported for ITT population (Open-Label and Randomized Phase), comprised of all participants who were randomized to LTG or placebo (only for Randomized Phase) and received at least one dose of the investigational product.
Groups:
- Open-Label and Open-Label Taper Phases: LTG: Participants (par.) received lamotrigine (LTG) up to a maximum dose depending on their age and concomitant bipolar medication group. Participants 10 -12 years of age received LTG up to a maximum dose of : 3 milligrams/kilograms (mg/kg)/day or 100 mg/day, whichever was less; or 6 mg/kg/day or 200 mg/day whichever was less; or 12 mg/kg/day or 300 mg/day whichever was less, depending on their bipolar medication group. Participants 13-17 years of age received LTG up to a maximum dose of 150 mg/day, 300 mg/day, or 400 mg/day depending on their bipolar medication group. Participants took LTG for a duration of up to 18 weeks. Participants discontinuing from the study during the Open-Label Phase entered an open Taper and Follow-up Phase.The Taper and Follow-up Phase may last up to 4 weeks, dependent on the dose of LTG the participant received during the Open-Label Phase.
- Randomized and Double-blind Taper Phases: Placebo: Participants received matching placebo in the evening for participants taking one dose and for participants taking two divided doses, one dose in the morning and one dose in the evening, for a duration of up to 36 weeks. Participants completing the Randomized Phase entered Double-Blind Taper and Follow-up Phase. The Taper and Follow-up Phase may last up to 4 weeks. The participant received Placebo during this Phase.
- Randomized and Double-blind Taper Phases: LTG: Participants received LTG equivalent to the dose established in the Open-Label Phase. Participants received LTG tablets in the evening for participants taking one dose and for participants taking two divided doses, one dose in the morning and one dose in the evening, for a duration of up to 36 weeks. Participants completing the Randomized Phase entered Double-Blind Taper and Follow-up Phase. The Taper and Follow-up Phase may last up to 4 weeks, dependent on the dose of LTG the participant received during the Randomized Phase.
Arm/Group | Open-Label and Open-Label Taper Phases: LTG | Randomized and Double-blind Taper Phases: Placebo | Randomized and Double-blind Taper Phases: LTG
Serious Adverse Events (participants affected / at risk) | 19/298 | 5/86 | 1/87
Other Adverse Events (participants affected / at risk) | 177/298 | 41/86 | 45/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label and Open-Label Taper Phases: LTG (N=298) | Randomized and Double-blind Taper Phases: Placebo (N=86) | Randomized and Double-blind Taper Phases: LTG (N=87)
Suicidal ideation (Psychiatric disorders) | 5 | 1 | 0
Agitation (Psychiatric disorders) | 3 | 0 | 0
Mania (Psychiatric disorders) | 3 | 1 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0
Impulsive behaviour (Psychiatric disorders) | 1 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0
Pressure of speech (Psychiatric disorders) | 1 | 0 | 0
Emotional disorder (Psychiatric disorders) | 0 | 0 | 1
Irritability (General disorders) | 2 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label and Open-Label Taper Phases: LTG (N=298) | Randomized and Double-blind Taper Phases: Placebo (N=86) | Randomized and Double-blind Taper Phases: LTG (N=87)
Headache (Nervous system disorders) | 106 | 18 | 18
Dizziness (Nervous system disorders) | 24 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 47 | 3 | 5
Nausea (Gastrointestinal disorders) | 39 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 23 | 0 | 0
Vomiting (Gastrointestinal disorders) | 25 | 3 | 5
Nasopharyngitis (Infections and infestations) | 25 | 5 | 7
Influenza (Infections and infestations) | 0 | 2 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 4 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 30 | 2 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 6
Insomnia (Psychiatric disorders) | 23 | 5 | 6
Suicidal ideation (Psychiatric disorders) | 16 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 5
Irritability (General disorders) | 16 | 14 | 7
Fatigue (General disorders) | 17 | 0 | 0
Pyrexia (General disorders) | 0 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.